CLINICAL TRIAL: NCT07306949
Title: A Multicenter, Open-Label, Single Arm, Post-Marketing Clinical Study to Evaluate the Therapeutic Effects of Acoramidis Hydrochlorideon Cardiac Biomarkers and Current Clinical Features in Patients With Transthyretin-type Cardiac Amyloidosis: The CARE ATTR Study
Brief Title: Real-Life Clinical Efficacy of Acoramidis in Participants With ATTR-CM and Association With Cardiac Biomarkers
Acronym: ATTR-CM
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Alexion Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: D9400L00001; 2025-RWE-000214 (Other: Alexion)
Record Dates: First submitted 2025-12-15; First posted 2025-12-29 (Actual); Last update posted 2026-01-07 (Actual); Status verified 2026-01

CONDITIONS: Transthyretin-type Cardiac Amyloidosis
Keywords: ATTR-CM; NT-proBNP; ODI; hs-cTnT; Acoramidis
MeSH Terms: interventions — attruby

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Acoramidis (Experimental): Participants will receive 800 mg of acoramidis twice daily for 18 months.
  Interventions: Drug: Acoramidis

INTERVENTIONS:
Drug: Acoramidis — Participants will receive acoramidis tablets orally.
  Other Names: acoramidis hydrochloride Byontra

SUMMARY:
The purpose of this study is to confirm that the treatment with acoramidis prevents the deterioration of the ATTR-CM disease progression index and that these indexes are surrogate markers of disease progression.

ELIGIBILITY:
Inclusion Criteria:

* Treatment history of ATTR-CM is one of the following:
* Naive participants: newly diagnosed with ATTR-CM and no prior treatment with drugs for ATTR-CM
* Switch participants: Participants who are using tafamidis, a TTR stabilizer, as treatment for ATTR-CM and who, in the judgment of the post-marketing clinical trial investigator (co-principal investigator), can be expected to benefit from switching to acoramidis.
* Naive participants must meet the following requirements:

  1. History of hospitalization for heart failure or heart failure symptoms requiring treatment, including diuretics
  2. Echocardiographic end-diastolic ventricular septal thickness greater than 12 millimeters (mm)
  3. Confirmed diagnosis of ATTR-CM (wild type or mutant) by one of the following diagnostic methods

     1. Tissue biopsy shows amyloid deposition and TTR precursor protein is identified by immunohistochemistry or mass spectrometry.
     2. Bone scintigraphy showing strong accumulation ** (Perugini score ≥ 2) consistent with myocardium and no M protein, negating the possibility of AL amyloidosis

Exclusion Criteria:

* Have confirmed diagnosis of AL amyloidosis
* Switch participants: prior treatment with gene silencing agents (pachysilane sodium, butrisilane sodium) as treatment for ATTR-CM (including when specifically scheduled to start treatment with a gene silencing agent)
* Likelihood of receiving a heart transplant within 1 year from the time screening begins
* Hypersensitivity to acoramidis, its metabolites, or additives in the formulation has been confirmed.
* Pregnant or lactating women
* Has a clinically significant medical condition, an abnormal laboratory test result, or a condition that may jeopardize the safety of the study participant, increase the risk of participation in the post-marketing clinical trial, or affect the study
* Participating in an interventional study other than this study, including a clinical trial
* In the opinion of the responsible (sub)physician for the post-marketing clinical trial, has a history of drug abuse, alcoholism, or psychiatric disorder that would preclude compliance with this Post-Marketing Clinical Study Protocol

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2025-10-01 (Actual); Primary Completion 2028-03-31 (Estimated); Study Completion 2028-03-31 (Estimated)

PRIMARY OUTCOMES:
Disease Progression Rate as Measured by N-terminal pro-brain-type Natriuretic Peptide (NT-proBNP) and/or Outpatient Diuretic Intensification (ODI) | Baseline through 12 months

SECONDARY OUTCOMES:
Disease Progression Rate as Measured by NT-proBNP and/or High-sensitivity Cardiac Troponin T (hs-CTnT) | Baseline through 12 months
Change from Baseline in Serum Transthyretin (TTR) | Baseline, 28 days
Number of Participants with a 30% Change from Baseline in NT-proBNP | Baseline, 12 months and 18 months
Change from Baseline in hs-CTnT | Baseline, 12 months and 18 months
Change from Baseline in Kansas City Cardiomyopathy Questionnaire (KCCQ-12) Overall Summary Score | Baseline, 12 months and 18 months
Change from Baseline in Estimated Glomerular Filtration Rate (eGFR) | Baseline, 12 months and 18 months

CONTACTS AND LOCATIONS:
Locations (15):
- Japan (15):
  - Research Site, Bunkyō City
  - Research Site, Kumamoto
  - Research Site, Kurume-shi
  - Research Site, Kyoto
  - Research Site, Mitaka-shi
  - Research Site, Nagoya
  - Research Site, Nankoku-shi
  - Research Site, Okayama
  - Research Site, Ōtsu
  - Research Site, Sagamihara-shi
  - Research Site, Sapporo
  - Research Site, Shinjuku-ku
  - Research Site, Suita-shi
  - Research Site, Tsu
  - Research Site, Yufu-shi

IPD SHARING:
Plan to Share IPD: Yes
Alexion has a public commitment to allow requests for access to study data and will be supplying a protocol, CSR, and plain language summaries.
Supporting Information: Study Protocol, SAP, CSR